CLINICAL TRIAL: NCT06435520
Title: Enhancing Hypnotic Medication Discontinuation in Primary Care Through Supervised Medication Tapering and Digital Cognitive Behavioral Insomnia Therapy
Brief Title: Enhancing Hypnotic Medication Discontinuation in Primary Care
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS4047
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-01

CONDITIONS: Insomnia; Hypnotic Dependence
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized trial to compare the combined digital cognitive behavioral therapy (dCBTI) / structured medication taper (SMT) intervention, to the SMT intervention delivered alone for producing hypnotic discontinuation and insomnia symptom improvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive behavioral therapy combined with structured medication tapering (Experimental): dCBTI delivered in tandem with SMT during intervention phase.
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy; Behavioral: Structured Medication Tapering
- Structured medication tapering alone (Experimental): Structured medication tapering delivered alone with general sleep hygiene information.
  Interventions: Behavioral: Structured Medication Tapering

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy — Adaptive cloud-based software delivering cognitive behavioral therapy tailored to the needs of the individual patient.
  Other Names: dCBTI; Sleepio
  Arms: Digital cognitive behavioral therapy combined with structured medication tapering
Behavioral: Structured Medication Tapering — A structured tapering of hypnotic (or other) medication to promote successful discontinuation by patients seeking to discontinue use.
  Other Names: SMT

SUMMARY:
Many individuals with insomnia seek treatment in primary care settings, where they often receive prescription hypnotic medications as their first and sometimes only treatment. However, extended use of these medications can lead to reliance and increased health risks, such as falls and cognitive impairments. While evidence-based approaches like physician-supervised medication tapering exist, they're not widely available in primary care.

Most primary care providers are willing to explore non-drug treatments like cognitive behavioral therapy for insomnia (CBTI), but accessing such treatments can be challenging outside of specialized sleep centers. This gap between research and practice underscores the need for cost-effective interventions to manage insomnia and help patients reduce their reliance on hypnotics in primary care.

In response to this need, the project aims to conduct a large randomized trial comparing a combined digital CBT (dCBTI) and medication tapering intervention with medication tapering alone. We'll recruit 430 patients reliant on hypnotics from 8-10 primary care clinics affiliated with the University of Colorado Medical School. The main goal is to assess the effectiveness of dCBTI+SMT compared to SMT alone in reducing hypnotic use and improving insomnia symptoms.

Additionally, we'll evaluate factors affecting the adoption and implementation of these interventions at the patient, provider, and system levels. This information will inform future implementation strategies to disseminate effective treatments in primary care.

Furthermore, we'll gather data to identify which patients benefit most from dCBTI+SMT. Overall, this study will provide valuable insights into the feasibility, clinical utility, and acceptability of these interventions in managing insomnia and reducing reliance on hypnotic medications in primary care. Ultimately, this project represents a crucial first step toward making accessible and cost-effective strategies available to improve the quality of life for millions of chronic users of sleep aids.

DETAILED DESCRIPTION:
Treatment-seeking insomnia sufferers most often present in primary care where their first and usually only treatment is a prescription hypnotic medication. More than 65% of individuals prescribed hypnotics use them for more than a year, and more than 30% remain on them for more than five years. Such agents may be useful for acute insomnia and certain cases with chronic sleep difficulties, but prolonged hypnotic use can lead to dependency and increased morbidity (e.g., falls, cognitive/driving impairments). Reducing or discontinuing hypnotics after prolonged use is a challenging task for both prescribing physicians and the patients who use them. Although evidenced-based physician-supervised medication tapering (SMT) protocols have shown efficacy, such interventions have yet to be disseminated widely in primary care. Most primary care providers (PCPs) are willing to refer their insomnia patients to alternative evidence-based non-drug treatments such as cognitive behavioral insomnia therapy (CBTI), but such treatment is often difficult to access outside of specialty sleep centers. Given this gap between research and clinical practice, there is a pressing need to develop and validate cost-effective interventions to facilitate the management of insomnia and hypnotic tapering in primary care. This study has been carefully designed to address these issues. Investigators will conduct a large randomized trial (RCT) to compare the combined digital CBT (dCBTI)/SMT intervention, to the SMT intervention delivered alone for producing hypnotic discontinuation and insomnia symptom improvement. A sample of 430 hypnotic-reliant patients drawn from 8-10 primary care clinics within a practice-based research network affiliated with the University of Colorado Medical School in Aurora, Colorado will serve as study participants. The main objective of the project is to compare the performance of dCBTI+SMT with SMT used alone for achieving hypnotic reduction/discontinuation and insomnia symptom improvement. In addition, investigators will incorporate an Effectiveness-Implementation assessment into the RCT to identify patient- provider- and system-level factors that may impact adoption, implementation and maintenance of the types of interventions tested. Findings from the effectiveness/implementation should help design future trials of implementation strategies identified herein to promote dissemination of dCBTI and SMT interventions into primary care should these treatments prove effective in the current trial. Investigators also will gather exploratory data to determine who responds best to dCBTI/SMT. This study will provide new and useful information about the feasibility, clinical utility, and patient-, provider-, and system-level acceptability of these interventions to manage insomnia and reduce/eliminate hypnotic use in primary care. This project should serve as a necessary first step toward the eventual dissemination of accessible, cost-effective strategies to manage a significant public health problem and improve the quality of life of millions of chronic users of controlled-substance sleep aids.

ELIGIBILITY:
Inclusion Criteria:

* a history of extended (> 6 consecutive months) and frequent (>5 nights/week on average) use of benzodiazepine (BZD) or non-BZD hypnotic medications;
* a desire to decrease/eliminate hypnotic use;
* a history of insomnia that meets DSM-560 criteria for insomnia disorder; and
* willingness to provide written informed consent to participate.

Exclusion Criteria:

* a lifetime diagnosis of any psychotic disorder, suicide attempts, or bipolar disorder;
* presence of an unstable, untreated, or terminal major medical or psychiatric disorder;
* alcohol or drug abuse within the past year;
* current use of a BZD for another disorder in addition to insomnia (e.g., seizure disorder, restless leg syndrome, anxiety disorder);
* pregnancy;
* significant cognitive impairment as suggested by a score of ≤ 24 on the Folstein Mini-Mental State Examination (MMSE);
* current use of medications known to cause insomnia (e.g., high dose corticosteroids);
* untreated comorbid sleep disorders;
* use of a sedating antidepressant or antipsychotic medication solely for sleep; and
* consuming >2 alcoholic beverages/day ≥5 times/week or any use of marijuana ≥5 times/week.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Hypnotic discontinuation rates | Post-treatment at weeks 22 and 49 of participation
  Rates of successful hypnotic discontinuation among participants
Insomnia remission rates | Post-treatment at weeks 22 and 49 of participation
  Rates of insomnia remission among participants

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Not planned.